# Family Champions Project Study Protocol Clinicaltrials.gov ID: NCT05298345 September 4, 2024

## Descriptive Evaluation Analysis Plan

## The Evaluation of the Family Champions Project in Dallas, TX

## A. Description of the intended intervention(s)

Anthem Strong Families' Family Champions Project (FCP) offers skill-building primary curriculum and support services to program participants. The evidence-based TYRO Leadership and TYRO Core Communication curricula, totaling 18 hours, are offered as group classes by trained facilitators in which low-income adults learn skills related to healthy relationships and financial wellbeing. Support services, including case management and additional, optional classes through Anthem's Mini-Clinic series, are available to all FCP participants.

The main intervention being tested in this descriptive evaluation is the multistep continuous quality improvement (CQI) cycle created by Midwest Evaluation and Research (MER) that aims to improve FCP program implementation. The content and components of each step in the process are described below.

# 1. <u>Step 1</u>: Real-Time Performance Assessment Reports (prepared and presented bi-weekly by evaluation lead and/or data manager)

- a. Report description use key indicators to track overall performance trends.
- b. Purpose
  - i. Provide real time monitoring of data entry and progress toward key metrics
  - ii. Familiarize CQI team staff with metrics that will be monitored and discussed throughout the lifetime of the project and in subsequent reports (Steps 2-5)
- c. Fidelity tracking number of CQI team meetings scheduled and held where Step 1 CQI reports are presented to the CQI team
- d. Dosage tracking -
  - i. Intended vs. actual amount received attendance of all CQI Team members at meetings for Step 1 Reports (i.e., number, names, roles) documented on CQI Team Tracking Sheet
- e. Performance Intervention Tracking CQI Tracking Sheet for Performance Issues and Interventions (ongoing entry and revision as needed)
- f. Feasibility Assessment
  - i. Focus on utility and user-friendliness of Step 1 report
  - ii. CQI Team Survey for Step 1: administered each program year to permanent staff on the CQI Team

# 2. <u>Step 2</u>: Performance Intervention Priorities Report (prepared and presented annually in quarter 2 of each grant year by evaluation lead)

- a. Report description compare overall performance trends by service site
- b. Purpose target improvement efforts by setting site-specific priorities for interventions
- c. Fidelity tracking
  - i. Intended amount of CQI to be offered based on intended report timeline
  - ii. Actual amount offered (# CQI Team meetings scheduled for Step 2 Reports on Outlook, # CQI Team meetings where Step 2 CQI Report was presented to CQI Team, # Step 2 reports created)

- d. Dosage tracking
  - i. Intended amount received attendance of all members at CQI Team meetings for Step 2 Reports (i.e., number, names, roles)
  - ii. Actual amount received CQI Tracking Sheet for Team Attendance (See AppendixB) for Step 2 Reports
- e. Feasibility Assessment
  - i. Focus on utility and user-friendliness of Step 2 report
  - ii. CQI Team Survey for Step 2: administered each program year to staff on the CQI Team
  - iii. Family Champions Project staff survey for Step 2: administered each program year to all frontline staff who help to develop targeted, site-specific interventions during staff meetings with leadership and with the CQI team on a rotating basis

# 3. <u>Step 3</u>: Performance Intervention Strategy Report (prepared for each service site in quarter 2 of each grant year by evaluation lead)

- a. Report description use key indicators to track performance trends for each site individually
- b. Purpose establish a performance intervention agenda for each site
- c. Fidelity tracking
  - i. Intended amount to be offered based on intended report timeline
  - ii. Actual amount offered (# CQI Team meetings scheduled on Outlook, # CQI Team meetings where Step 3 CQI Report presented to CQI Team, # Step 3 reports created)
- d. Dosage tracking
  - i. Intended amount received attendance of all members at CQI Team meetings for Step 3 Reports (i.e., number, names, roles)
  - ii. Actual amount received CQI Tracking Sheet for Team Attendance for Step 3 Reports
- e. Feasibility assessment
  - i. Focus on utility and user-friendliness of Step 3 report
  - ii. CQI Team Survey for Step 3: administered each program year to staff on the CQI Team

# 4. <u>Step 4</u>: Performance Intervention Results Reports (prepared annually in quarter 4 of each grant year by evaluation lead)

- a. Report description examine performance trends before and after an intervention at each site, looking for improvements and comparing to the relevant standards
- b. Purpose assess results of interventions on performance outputs to determine whether improvements were made for the relevant standard
- c. Fidelity tracking
  - i. Intended amount to be offered based on intended report timeline
  - ii. Actual amount offered (# CQI Team meetings scheduled on Outlook, # CQI Team meetings where Step 4 CQI Report presented to CQI Team, # Step 4 reports created)
- d. Dosage tracking
  - i. Intended amount received attendance of all members at CQI Team meetings for Step 4 Reports (i.e., number, names, roles)

- ii. Actual amount received CQI Tracking Sheet for Team Attendance for Step 4 Reports
- e. Feasibility assessment
  - i. Focus on utility and user-friendliness of Step 4 report
  - ii. CQI Team Survey for Step 4: administered each program year to staff on the CQI Team
  - iii. FCP Staff Survey for Step 4: administered each program year to all frontline staff who develop performance interventions with the CQI team

**Table 1**. Description of intended intervention components, content, dosage and implementation schedule, delivery, and focal populations

| Components | Content | Dosage and schedule | Delivery | Focal population |
|---|---|---|---|---|
| CQI Process Step 1 | Monitoring overall and recent program performance using nFORM operational reports, local evaluation survey data, and the query tool | Reports are prepared<br>bi-weekly and<br>discussed at bi-weekly,<br>hour-long CQI team<br>meetings | Virtual CQI team meetings are held bi-<br>weekly on Tuesday mornings; the evaluation lead facilitates meetings, and Step 1 reports are presented by the evaluation lead and/or data manager | CQI team members<br>(program director,<br>program manager,<br>evaluation lead, data<br>manager(s)) |
| CQI Process Step 2 | Monitoring the same performance metrics as presented in the Step 1 report, but broken down by service site using nFORM operational reports, local evaluation survey data, and the query tool | Reports are prepared annually in the second quarter of each grant year and discussed at standing CQI team meetings and program staff meetings | Existing CQI team meetings are used to present and discuss Step 2 report findings; the evaluation lead facilitates the meetings and presents the Step 2 reports to the CQI team. Following the CQI team discussion, program leadership shares the Step 2 report findings with front line staff during staff meetings to solicit ideas for interventions | CQI team members (program director, program manager, evaluation lead, data manager(s); rotating front line staff member); Anthem program staff (case managers, facilitators, recruitment and retention specialists) who work at the sites being discussed in the Step 2 reports |
| CQI Process Step 3 | Offering the same conclusions as the Step 2 report but focusing on one service site per Step 3 report; uses nFORM operational reports, local evaluation survey data, and the query tool | Reports are prepared annually in the second quarter of each grant year and discussed at standing CQI team meetings | Step 3 reports are<br>sent to the program<br>director who<br>distributes each site's<br>Step 3 report to the<br>relevant program staff<br>who work at that site | CQI team members<br>(program director,<br>program manager,<br>evaluation lead, data<br>manager(s)); program<br>staff for specific sites<br>(case managers,<br>facilitators) |

| Components | Content | Dosage and schedule | Delivery | Focal population |
|---|---|---|---|---|
| CQI Process Step 4 | Assessing the results of targeted interventions that were put in place at specific sites based on the findings of the Step 2 and Step 3 reports | Reports are prepared annually in the fourth quarter of each grant year and discussed at standing CQI team meetings | Existing CQI team meetings are used to present and discuss Step 4 report findings (e.g., did the targeted metrics improve after implementing interventions? Does the metric now meet relevant standards? Were there any challenges with the implementation of interventions? How did frontline staff, leadership, and facility staff find the intervention?); the evaluation lead facilitates the CQI team meetings and presents the Step 4 reports to the CQI team. Program leadership share Step 4 report findings with frontline staff in staff meetings. | CQI team members (program director, program manager, evaluation lead, data manager(s)); program staff (case managers, facilitators, recruitment and retention specialists) who are able to 1) provide feedback on challenges and successes with the implementation of the intended intervention, 2) see the results of the intervention |
| Relationship skills<br>workshops | Healthy relationships<br>curriculum (TYRO<br>Core Communication;<br>TYRO Leadership) | A total of 18 hours,<br>with six two-hour<br>sessions occurring<br>weekly (TYRO<br>Leadership) plus two<br>three-hour sessions<br>occurring weekly<br>(TYRO Core<br>Communication) | Group lessons provided online via Zoom or in-person at service sites; two trained facilitators lead every session | Individuals in the<br>greater Dallas-Fort<br>Worth area with low<br>income |

**Table 2**. Staff education and training (initial and ongoing)

| Component | Education and initial training | Ongoing training |
|---|---|---|
| Relationship skills<br>workshop | All facilitators, case managers, intake specialists, and other members of the staff must complete the workshop as a participant before entering the certified TYRO Facilitator training component. Once the training is complete, each facilitator observes an experienced staff | Facilitators complete an annual refresher process to ensure curriculum fidelity. That process includes observations by the Program Manager, Program Director, or another qualified designee. We attempt to provide opportunities to become recertified every two to three years. Other |

| Component | Education and initial training | Ongoing training |
|---|---|---|
| | prior to undergoing observation of their group facilitation. Once completed, they are considered a certified TYRO curriculum facilitator. | facilitation or case management training is offered through targeted webinars or staff development sessions. |
| CQI process | At the beginning of the grant cycle, Anthem held a 3-day training to discuss the specifics of the grant and evaluation, and the purpose and process of CQI were discussed in detail at this initial training. As new staff are onboarded, they receive an explanation of the purpose and process of CQI, both from program leadership and from more experienced staff. | The purpose and process of CQI is reinforced on an ongoing basis. Starting with more experienced staff who fully understand their day-to-day roles, frontline staff are invited to sit in on CQI team meetings on a quarterly rotating basis to help them understand the value of the CQI process and how their role fits into the larger picture. CQI report findings are discussed with staff at weekly staff meetings. |

## **B.** Outcomes study

This section describes the research questions, evaluation enrollment process, data collection procedures, outcome measures, and analytic approach for the outcomes study.

#### 1. Research questions

RQ1.1: Did the multistep CQI process support changes in primary workshop dosage, program attrition rates, or survey response rates at the <u>program</u> level?

RQ2: Did meaningful improvements in primary workshop dosage, survey response rates, or program attrition rates vary by service site for sites that focused on improving the same metrics?

RQ3 [secondary]: Do participants report healthier partner relationship attitude outcomes after program participation, as compared to baseline?

RQ4 [secondary]: Was level of dosage associated with reporting heathier partner relationship attitude outcomes after program participation, as compared to baseline?

#### 2. Outcomes evaluation enrollment

This study was initially approved by Solutions IRB on 03/29/2021 and has been annually reviewed and approved on 03/15/2022, 03/07/2023, and 3/11/2024. Additionally, revisions to the study were submitted as amendments and were approved on 05/17/2022, 02/15/2023, and 08/29/2023.

Participants for the program, and thus the study, are recruited primarily from community partnerships, walk-ins to Anthem Strong Families, radio and social media advertising, and word of mouth referrals.

Program service locations have varied throughout the implementation of the program but have included:

- Schools
  - Stephen C. Foster Elementary School
  - Herbert Marcus Elementary School
  - Burnet Elementary School
- Treatment Centers / Transitional Facilities
  - Soul's Harbor Treatment Center
  - Free Man House Transitional Living Facility
  - Shurrun's House Sober Living Facility
  - Gateway Foundation Treatment Center
- Vickery Meadow Youth Development Foundation
- Buckner Children and Family Services, Family Hope Center at Bachman Lake
- Virtual services provided via Zoom

The projected enrollment and desired sample size for the study is 800 participants. The final report will include a breakdown of the number of sites, number of staff at each site, and number of participants at each site.

To be eligible for the program, and thus the study, participants must be 1) low-income individuals, 2) at least 18 years of age, 3) with no open criminal cases (can be deferred), and 4) able to speak and understand English or Spanish.

Consent for enrollment into the evaluation happens during program orientation, prior to the start of the first primary workshop. A consent form is provided to participants, and a script is read by either the facilitator or the data manager, explaining the study activities and the potential risks and benefits. Participants sign and date the consent form and return it to the data manager, who logs the record in a consent spreadsheet on MER's secure Dropbox.

Enrollment into the study began April 22, 2021 and is estimated to conclude February 15, 2025.

#### 3. Data sources and data collection

The data source for the program implementation and performance outcome measures is nFORM administrative data. Program staff are responsible for entering and updating client and workshop information, including workshop attendance and current client status, on an ongoing basis. These data are summarized bi-weekly in Step 1 CQI reports with metrics at the program level and annually in Step 2-4 CQI reports with metrics at the site level to monitor trends in program enrollment, workshop dosage, program attrition rates, and survey response rates.

The data source for participant outcomes related to healthy partner relationship attitudes is the nFORM

Healthy Marriage Adult Program survey, administered at orientation before the first primary workshop (entrance survey) and at the final primary workshop session (exit survey).

**Table 3**. Sources of data to address the research questions

| Data source | Timing of data collection | Mode of data collection | Start and end date of data collection |
|---|---|---|---|
| nFORM<br>administrative data | Ongoing | Program staff enter and update data related to enrollment, attendance, and client status | Start: April 2021<br>End: April 2025 |
| nFORM Healthy<br>Marriage Adult<br>Program Survey | At orientation before the first primary workshop (entrance survey) and at the end of the final primary workshop session (exit survey) | Online via tablet or on paper as necessary | Start: April 2021<br>End: April 2025 |

#### 4. Outcome measures

The main outcomes of interest addressed by the multistep CQI process are primary workshop dosage, participant attrition rates, and nFORM survey response rates, as these are key program performance metrics with targets set by the federal funders. The first research question looks at changes in each of these metrics over time overall across all service sites (program level), and the second research question looks at changes in each of these metrics over time broken down by service site for sites that focused on the same metrics. This will involve an assessment of any changes in metrics after intervention strategies were implemented, including whether performance targets were reached and whether improvements were meaningfully large. Potential ceiling and floor effects are mitigated during the process of selecting which metrics to attempt to improve via intervention strategies (i.e., metrics that are already at or close to targets are not selected for intervention); however, potential ceiling and floor effects will also be addressed by providing baseline data for metrics targeted for interventions at each service site.

The secondary research questions about participant-level attitude changes after program participation are assessed by constructing a composite measure calculated as the average of five nFORM survey items related to partner trust and intimacy. If more than one survey item within the composite is missing for a respondent, the value of the outcome measure will be set to missing.

**Table 4**. Outcomes used to answer the research questions

| Research question | Outcome name | Description of the outcome measure | Source of the measure | Timing of measure |
|---|---|---|---|---|
| RQ1 | Dosage | The outcome measure is the percent of target primary workshop hours received by program participants | nFORM operational<br>report: Primary<br>Workshop<br>Participation Detail | Attendance is recorded after each workshop session |
| RQ1 | Attrition | The outcome measure is the percent of program participants who leave the program without completing at least 90% of primary workshop hours | nFORM operational<br>report: Client Status<br>Summary | Ongoing |

| Research question | Outcome name | Description of the outcome measure | Source of the measure | Timing of measure |
|---|---|---|---|---|
| RQ1 | Survey response rates | The outcome measure is the percent of eligible participants who completed nFORM entrance and exit surveys | nFORM operational<br>report: Survey<br>Completion<br>Summary | Ongoing |
| RQ2 | Dosage | The outcome measure is the percent of target primary workshop hours received by program participants at each service site | nFORM operational<br>report: Primary<br>Workshop<br>Participation Detail | Attendance is recorded after each workshop session |
| RQ2 | Attrition | The outcome measure is the percent of program participants who leave the program without completing at least 90% of primary workshop hours at each service site | nFORM operational<br>report: Client Status<br>Summary | Ongoing |
| RQ2 | Survey response rates | The outcome measure is the percent of eligible participants who completed nFORM entrance and exit surveys at each service site | nFORM operational<br>report: Survey<br>Completion<br>Summary | Ongoing |
| RQ3 | Healthy partner relationship attitudes | The outcome measure is a scale (value range 1-5) calculated as the average of five survey items measuring trust and intimacy | nFORM Healthy<br>Marriage Adult<br>Program survey<br>D10.a-e (entrance<br>and exit) | During orientation<br>(entrance) and after<br>the final workshop<br>session (exit) |
| RQ4 | Healthy partner relationship attitudes | The outcome measure is a scale (value range 1-5) calculated as the average of five survey items measuring trust and intimacy | nFORM Healthy<br>Marriage Adult<br>Program survey<br>D10.a-e (entrance<br>and exit) | During orientation<br>(entrance) and after<br>the final workshop<br>session (exit) |

## A. Implementation study

This section describes the research questions, the data used to answer the research questions, and the methods used to analyze the data and describe the findings of the process or implementation study.

#### 1. Research questions

The research questions for this implementation study relate to fidelity to, and engagement with, the planned multistep CQI process. The implementation study seeks to understand how closely the CQI process followed the original outlined plan and how understandable, useful, and engaging program staff found each step of the CQI process. Additionally, the implementation study seeks to understand what contextual factors affected the implementation of the multistep CQI process and to identify best practices and lessons learned about implementing a CQI process that could be shared with the broader field.

**Table 5**. Research questions for each implementation element

| Implementation element | Research question |
|---|---|
| Fidelity | To what extent were the five steps of the CQI process carried out as intended each grant year? |
| | What were the unplanned adaptations to the key CQI process components? |

| Implementation element | Research question |
|---|---|
| Engagement | How understandable did CQI team members, and program staff broadly for Step 2 and Step 4, find the reports for each step of the CQI process? |
| | How engaged were CQI team members and program staff in each step of the CQI process? |
| Context | How well did the implementation of the multistep CQI process go for program and evaluation staff? |
| | What external events affected the implementation of the multistep CQI process? |
| | What are some best practices and lessons learned for improving the multistep CQI process? |

#### 2. Implementation evaluation enrollment

The implementation study was initially approved along with the outcome study by Solutions IRB on 03/29/2021 and has been annually reviewed and approved three times on 03/15/2022, 03/07/2023, and 3/11/2024. Additionally, revisions to the study were submitted as amendments and were approved on 05/17/2022, 02/15/2023, and 08/29/2023.

The sample for the implementation evaluation is made up of staff from Anthem Strong Families. The final report will include information about staff demographics, role types, and participation levels. Permanent members of the CQI team are surveyed after each step of the CQI process has been completed, and the program staff more broadly are surveyed after reviewing Step 2, 3, and 4 reports that are relevant to the service sites where they work with participants. Staff are also interviewed during annual site visits.

Because the data sources for the implementation evaluation are staff satisfaction surveys that are not administered to program participants, no consent is collected, and no incentives are offered for survey completion.

#### 3. Data sources and data collection

The data sources for the implementation evaluation are CQI process tracking logs (See Appendix C), staff satisfaction surveys administered on Qualtrics (see Appendix A), and staff interviews.

The evaluation lead and data manager from Midwest Evaluation and Research are responsible for tracking and logging the delivery of interventions and reports that are associated with each step of the multistep CQI process. When program staff decide on a targeted intervention to implement at a given site, evaluators document when (with which cohort, or on which specific date) and where (which service site or sites) the intervention is being put into place. The date that each CQI report is delivered is also documented. Additionally, CQI meeting attendance is tracked on an ongoing basis after each bi-weekly meeting to assess CQI team engagement with the process.

The evaluation lead is responsible for creating and administering staff satisfaction surveys for each step of the multistep CQI process. After reviewing Step 2, 3, and 4 reports annually with the CQI team, anonymous satisfaction surveys are delivered to CQI team members by the evaluation lead using an anonymous Qualtrics link via email. Although Step 1 reports are delivered bi-weekly to CQI team members, satisfaction surveys for the Step 1 reports are sent out annually. After the Program Director presents Step 2 and Step 4 annual reports with relevant program staff during staff meetings, an anonymous satisfaction survey is sent

to staff members using an anonymous Qualtrics link via email. Satisfaction survey instruments can be found in Appendix A.

Additionally, staff interviews during annual site visits provide more information about lessons learned, best practices, how CQI findings are being applied to program implementation, and suggestions for improving the CQI multistep process. MER evaluation staff will also reflect at the end of the project on successes and challenges related to the implementation of the multistep CQI process to inform future CQI efforts.

**Table 6**. Data for addressing the implementation research questions

| <del>-</del> | | | | _ |
|---|---|---|---|---|
| Implementation element | Research question | Data source | Timing and frequency of data collection | Party responsible for data collection |
| Fidelity | To what extent were the five steps of the CQI process carried out as intended each grant year? | CQI process tracking log<br>(See Appendix C) | Updated after each step<br>of a CQI cycle | Evaluation lead and/or<br>data manager |
| Fidelity | What were the unplanned adaptations to key CQI process components? | CQI process tracking log<br>(See Appendix C) | Ad hoc | Evaluation lead and/or data manager |
| Engagement | How understandable did CQI team members, and program staff broadly for Step 2 and Step 4, find the reports for each step of the CQI process? | CQI team satisfaction<br>surveys; staff<br>satisfaction surveys<br>(See Appendix A) | Annually after the completion of each step of the CQI process has been completed | Evaluation lead |
| Engagement | How engaged were CQI team members and program staff in each step of the CQI process? | CQI team satisfaction<br>surveys; staff<br>satisfaction surveys<br>(See Appendix A) | Annually after the completion of each step of the CQI process has been completed | Evaluation lead and/or data manager |
| Engagement | How engaged were CQI team members in meetings? | CQI team meeting<br>attendance logs (See<br>Appendix B) | Bi-weekly after each<br>CQI team meeting | Evaluation lead |
| Context | How well did the implementation of the multistep CQI process go for program and evaluation staff? | Staff interviews;<br>evaluator retrospective | Annually during site visits | Evaluation staff |
| Context | What external events affected the implementation of the multistep CQI process? | Staff interviews;<br>evaluator retrospective | Annually during site visits | Evaluation staff |

| Implementation element | Research question | Data source | Timing and frequency of data collection | Party responsible for data collection |
|---|---|---|---|---|
| Context | What are some best practices and lessons learned for improving the multistep CQI process? | Staff interviews;<br>evaluator retrospective | Annually during site visits | Evaluation staff |